CLINICAL TRIAL: NCT05901116
Title: The Efficacy of Serratus Posterior Superior Intercostal Plane Block (SPSIPB) on Postoperative Pain and Total Analgesic Consumption in Patients Undergoing Reduction Mammoplasty Surgery: Case Series
Brief Title: The Efficacy of SPSIPB on Postoperative Pain in Patients Undergoing Reduction Mammoplasty Surgery: Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Assisstant Professor, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPSIPB on mammoplasty
Record Dates: First submitted 2023-06-01; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain
Keywords: serratus posterior superior intercostal plane block; postoperative pain; reduction mammoplasty; regional anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPSIPB (Other): SPSIPB is the intervention used in this study. It was performed when the patient is in lateral decubitis position. A high frequency (7-12 MHz) linear transducer of the ultrasound device is placed at the spinae scapula level in the transverse plane, and the upper medial border of the scapula, the trapezius muscle, rhomboid muscle, serratus posterior superior muscle (SPSM) and the second and third ribs are visualized. The sonovisible needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs in order to reach the fascial plane between the SPSM and intercostal muscles. After contact of the needle with the rib gently, 1-2mL of saline is used to confirm the correct plane, and a total of 30 mL of 0.25% bupivacaine is administered to the superficial to the intercostal muscle. Tramadol (intravenous analgesic drug) at a concentration of 4 mg per 1 ml was administered with patient-controlled analgesia (PCA) device (max dose: 400 mg /day)
  Interventions: Other: Serratus posterior superior intercostal plane block (SPSIPB)

INTERVENTIONS:
Other: Serratus posterior superior intercostal plane block (SPSIPB) — Serratus posterior superior intercostal plane block is the intervention used in this study. It was performed when the patient is in lateral decubitis position. A high frequency (7-12 MHz) linear transducer of the ultrasound device is placed at the spinae scapula level in the transverse plane, and the upper medial border of the scapula, the trapezius muscle, rhomboid muscle, serratus posterior superior muscle (SPSM) and the second and third ribs are visualized. The sonovisible needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs in order to reach the fascial plane between the SPSM and intercostal muscles. After contact of the needle with the rib gently, 1-2mL of saline is used to confirm the correct plane, and a total of 30 mL of 0.25% bupivacaine is administered to the superficial to the intercostal muscle.

SUMMARY:
The aim of this study is to investigate the postoperative analgesic efficacy of SPSIPB and its effect on opioid consumption in patients undergoing reduction mammoplasty.

DETAILED DESCRIPTION:
Ten patients had serratus posterior superior intercostal plane block (SPSIPB) as the intervention. Patients had SPSIPB with 0.25% bupivacaine (total volume of 30 ml) before the surgery in operating room. Numerical rating scale (NRS) was used to assess postoperative pain on 1st, 6th, 12th and 24th hour after the surgery. Total tramadol consumption was calculated by using patient-controlled analgesia (PCA) device. Patient satisfaction was assessed by using quality of recovery-15 (QoR15) scale. Paracetamol was planned as resque analgesic drug (maximum dose: 3 gr/day).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who underwent reduction mammoplasty under general anesthesia and are American Society of Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* Patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) scores | Postoperative 24 hours
  Numerical rating scale was used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.
Total Tramadol consumption | Postoperative 24 hours
  Postoperative analgesic (tramadol) need was measured by using patient-controlled analgesia (PCA) device.

SECONDARY OUTCOMES:
Resque analgesic need | Postoperative 24 hours
  Total paracetamol need was recorded as "milligram" in unit despite of tramadol administration.
Quality of Recovery scores | Postoperative 24 hours
  Quality of recovery-15 (QoR15) scale was used for the assessment of patients satisfaction. The scores of QoR15 changes between 0 to 150 points. 0 point means "there is no satisfaction." Higher scores mean indicating a good quality of recovery and better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093